CLINICAL TRIAL: NCT06554691
Title: Exploring the Immunological Basis in the Evolution of Tree Nut and Peanut Allergy During Treatment Care for Understanding Markers and Treatment Targets
Brief Title: Understanding the Immune System's Role in Tree Nut and Peanut Allergies: Key Biomarkers for Diagnosis and Treatment Monitoring and Treatment Targets
Acronym: Markers4Care
Status: Active, not recruiting | Type: Observational
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor
Other Study IDs: 230043_Markers4Care; PRIDE 19/14254520 i2TRON (Other Grant/Funding Number: Luxembourg National Research Fund); PRIDE 16749720 NEXTIMMUNE2 (Other Grant/Funding Number: Luxembourg National Research Fund)
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Food Allergy; Food Allergy in Children; Food Allergy Peanut; Tree Nut Allergies; Allergy;Food; Oral Immunotherapy for Food Allergy
Keywords: food allergy; peanut allergy; tree nut allergy; nut allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Nut Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — Biological samples: Whole blood, sera, plasma and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Immunotherapy: Participants in this group undergo oral immunotherapy as part of their routine management of their nut allergies
- Avoidance diet: Participants in this group are on strict avoidance diet as part of their nut allergy management

SUMMARY:
Peanut and tree nuts belong to the main elicitors of pediatric food allergy and are the main cause of near fatal reactions in children requiring emergency management. Oral immunotherapy has emerged as an alternative treatment option for the management of food allergies, to enhance patients' safety and quality of life. Monitoring if the therapy is working relies on oral food challenges during the course of treatment. There is a clear need for reliable biomarkers that are reflective of the clinical progression during oral food challenges and during immunotherapy that would help with patient stratification and possibly for personalized treatment approaches in the future

The aim of this study is to measure immune parameters in the blood of nut-allergic participants during oral food challenges and during the course of oral immunotherapy.

The main questions the study aims to answer are:

1. Identify immune markers that correlate with clinical reactivity
2. Identify immune changes and markers that correlate with immunotherapy outcome

Researchers will compare these immune parameters between nut-allergic participants on oral immunotherapy and with nut-allergic participants on avoidance diet. Additionally, we will also compare the immune parameters of these nut-allergic participants with those healthy adults.

DETAILED DESCRIPTION:
Background: The prevalence of peanut together with tree nut allergies have increase over the years and accounts for most of the life-threatening reactions even to minute doses of the allergen. Consequently, peanut and tree-nut allergies cause significant physical and mental burden to patients and their caretakers due to anxiety and fear of anaphylaxis from accidental exposures, stress from following a strict elimination diet, lack of proactive management plan and due to the low probability of natural recovery of such allergies. For decades, the management relied on a strict avoidance of the culprit foods. Oral immune therapy (OIT) is a ground breaking alternative modality to strict avoidance diets. OIT consist of gradual introduction of low doses of the implicated food allergen with the aim to modulate the patient's immune response and help build immunological and clinical tolerance. Though OIT has its strong advantages, the clinical outcome is variable among the patients. Therefore, there is a clear need for reliable ex-vivo biomarkers that are reflective of the clinical progression and therapy outcome that could aid with a more accurate patient stratification for personalized treatment approaches in the future.

Aims: This project aims at measuring immune targets, antibodies, immune cells and immune mediators, in patients' blood during oral food challenges (OFCs) and during the course of standard-of-care oral immunotherapy to identify new immune markers correlating to with the clinical outcome of the treatment. The identification of immune modifications during OIT will allow us to endotype patients and possibly aid in unraveling markers of food challenges and therapy progression as well as OIT outcome.

Luxembourg partners: The Luxembourg Institute of Health (LIH), Department of Infection and Immunity (DII; head Prof. M. Ollert) has the scientific project lead (Principal Investigator Dr. A. Kuehn). Main clinical partners are Dr. F. Codreanu-Morel and Dr. V. Petit-Cordebar from the National Unit of Immunology-Allergology, Centre Hospitalier (CHL), Luxembourg. Medical Principal Investigator for healthy controls is Dr. Alessia Pochesci, MD, Clinical and Epidemiological Investigation Center (CIEC), Luxembourg Institute of Health (LIH), Luxembourg. The Integrated Biobank of Luxembourg (IBBL) will prepare and store a subset of clinical samples until use. Other biological samples are prepared and stored at DII, LIH. Clinical samples (blood, sera, plasma,stool) will be analyzed at DII, LIH.

Project implementation: The clinicians at CHL will perform detailed clinical examinations of participants including skin prick test (SPT), serological analysis for specific IgE and food challenges to the implicated food allergen as per their routine clinical practice at the National Unit of Immunology-Allergology (CHL). Based on the European Academy of Allergy and Clinical Immunology (EAACI) guidelines and procedures established at CHL, all peanut- and tree-nut-allergic participants eligible for the study will undergo a baseline OFC. OFC is adapted from PRACTALL protocol and allergen doses are adjusted according to the clinical reactivity of the patient.

For participants eligible for immunotherapy (N= 30 Peanut-OIT and N=30 Tree nut-OIT), the OIT is based on the established protocol at the clinic and adapted from the current literature. Briefly, participant ingest incremental doses of the allergen (peanut/tree nut) at home until they reach a maintenance dose of 300 mg nut-protein in approximately 26 weeks (6 months). This initial phase of OIT is termed as the build-up phase. This is then followed by continued daily intake of this maintenance dose. After a minimum of 12 months of the maintenance phase of OIT, participants undergo another final OFC at the hospital to assess for desensitization to peanut or tree nut. Participants follow up at the hospital every 6 months i.e at end of the build-up phase, after 6 months and after 12 months of daily intake of maintenance dose.

Participants who are not eligible for OIT (N=30 peanut and tree-nut allergic) and who are on avoidance diet, are also followed up every 6 months for 18 months. However, final OFC will not be done for these participants.

The data collection of the study participants is carried out by the medical lead.

In addition, healthy adults (N=20) tolerating any type of nut and without any known food allergies will be recruited as controls. Dr. Alessia Pochesci, CIEC, LIH is responsible for the data collection from these healthy participants.

Blood sample collection:

i) For OIT group:

* During the baseline and final OFC , blood samples will be collected at the beginning, during and at the end of the food challenge in three different vials.
* During OIT follow-up, a one-time blood sample will be collected at the end of the build-up phase and after 6 months of maintenance phase in addition to the routine blood collection during these follow-up visits.

ii) For avoidance group:

* During the baseline OFC , blood samples will be collected at the beginning, during and at the end of the food challenge.
* During follow-up visits, one-time blood sampling will be taken six monthly i.e. at 6, 12 and 18 months after the baseline OFC.

iii) Healthy Adult participants: A one-time blood sampling will be done.

Stool sample collection:

Stool sample will be collected from nut-allergic participants at baseline and after the completion of a minimum of 18 months of the study duration using commercial at-home stool sampling kits. Participants receive a collection kit, containing special sampling tubes, accessories and instructions.

Collected clinical samples will be pseudonymized at the clinical centers. A synonym list containing the information on the identify of the participants recruited and their corresponding pseudonym, will be available at the clinical center only (medical investigators). Personal data is protected under the regulation (EU) 2016/679 of 27 April 2016 on the protection of individuals with regard to the processing of personal data (GDPR) and the law of 1 August 2018 on the organization of the National Data Protection Commission and the General Data Protection Act.

ELIGIBILITY:
For Peanut and Tree nut Allergic participants

Inclusion criteria:

* More than 2 years
* Male or Female
* Allergic to peanut (assessed by anamnesis, skin reactivity testing, sera testing for specific IgE)
* Sign an Informed Consent

Exclusion criteria:

* Pregnancy
* Less than 2 years of age
* Co-existing chronic medical condition such as cardiovascular disorders
* Peanut or tree nut-allergic patients/families who are unwilling to undergo oral food challenges

The eligible participants will be assigned to the oral immunotherapy (OIT) group but if they are not eligible for OIT based on either on the reasons mentioned below, they will be assigned to the avoidance group.

Reasons for ineligibility of OIT :

* risk of poor compliance with immunotherapy
* lack of understanding of the OIT protocol
* uncontrolled asthma
* incompatibility with lifestyle (regular intense physical activities, multiple vacations)
* unwilling to undergo OIT
* long-term or frequent use of non-steroidal anti-inflammatory drugs
* multiple nut allergy with no direct clinical benefit of OIT to one nut
* co-existing comorbidities such as active systemic autoimmune diseases, active malignancy, eosinophilic esophagitis.

For Healthy Controls

Inclusion Criteria:

* Adults
* Male or Female
* Sign an Informed Consent
* Tolerates any type of nut
* No known food allergy

Exclusion Criteria:

* Pregnancy
* Co-existing chronic medical condition such as cardiovascular disorders

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For peanut and tree nut-allergic cohort, participants are selected from the Immnulogy and Allergology Deparment at the Centre Hospitalier de Luxembourg.
  For the healthy adults cohort, participants are recruited from the Luxembourg population.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Baseline Immunophenotyping of peanut versus tree nut allergic participants | From enrollment to after 18 months of oral immunotherapy
  To identify the baseline immuonophenotypes using mass cytometry/flow cytometry for peanut versus tree nut-allergic participants and to correlate these findings with the oral food challenge and oral immunotherapy outcome.
Immune changes during Oral Food Challenge and Immune changes from baseline to 18 months of Oral Immunotherapy | From enrollment to after 18 months of immunotherapy (for oral immunotherapy group) and from enrollment to the end of 18 months follow up for avoidance diet group
  To investigate and map immune changes reflective of inflammation and cell migration during oral food challenge (OFC) and oral immunotherapy (OIT) in children with nut allergy. We will compare the immune profiles from OFC samples before commencing OIT vs OFC after 18 months of OIT. The immnue changes will also be compared to those nut-allergic participants on avoidance diet.

SECONDARY OUTCOMES:
Integration of the immune cell changes observed from the primary outcome with the serological and other immunological parameters | From enrollment to the end of 18 months of immunotherapy (for oral immunotherapy group) and to the end of 18 months follow up (for the avoidance group)
  Serological parameters such as specific IgE and immune mediators such as cytokines measured at baseline and follow up visits will be correlated with the immune cell changes observed from the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Annette Kuehn, Principal Investigator — Luxembourg Institute of Health
Locations (2):
- Luxembourg (2):
  - Centre Hospitalier de Luxembourg, Luxembourg
  - Clinical and Epidemiological Investigation Center, Luxembourg Institute of Health, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luce S, Chinthrajah S, Lyu SC, Nadeau KC, Mascarell L. Th2A and Th17 cell frequencies and regulatory markers as follow-up biomarker candidates for successful multifood oral immunotherapy. Allergy. 2020 Jun;75(6):1513-1516. doi: 10.1111/all.14180. Epub 2020 Jan 31. No abstract available. PMID 31930521
- [Background] Bajzik V, DeBerg HA, Garabatos N, Rust BJ, Obrien KK, Nguyen QA, O'Rourke C, Smith A, Walker AH, Quinn C, Gersuk VH, Farrington M, Jeong D, Vickery BP, Adelman DC, Wambre E. Oral desensitization therapy for peanut allergy induces dynamic changes in peanut-specific immune responses. Allergy. 2022 Aug;77(8):2534-2548. doi: 10.1111/all.15276. Epub 2022 Mar 14. PMID 35266148
- [Background] Monian B, Tu AA, Ruiter B, Morgan DM, Petrossian PM, Smith NP, Gierahn TM, Ginder JH, Shreffler WG, Love JC. Peanut oral immunotherapy differentially suppresses clonally distinct subsets of T helper cells. J Clin Invest. 2022 Jan 18;132(2):e150634. doi: 10.1172/JCI150634. PMID 34813505
- [Background] Santos AF, Du Toit G, O'Rourke C, Becares N, Couto-Francisco N, Radulovic S, Khaleva E, Basting M, Harris KM, Larson D, Sayre P, Plaut M, Roberts G, Bahnson HT, Lack G. Biomarkers of severity and threshold of allergic reactions during oral peanut challenges. J Allergy Clin Immunol. 2020 Aug;146(2):344-355. doi: 10.1016/j.jaci.2020.03.035. Epub 2020 Apr 18. PMID 32311390
- [Background] Calise J, DeBerg H, Garabatos N, Khosa S, Bajzik V, Calderon LB, Aldridge K, Rosasco M, Ferslew BC, Zhu T, Smulders R, Wheatley LM, Laidlaw TM, Qin T, Chichili GR, Adelman DC, Farrington M, Robinson D, Jeong D, Jones SM, Sanda S, Larson D, Kwok WW, Baloh C, Nepom GT, Wambre E; IMPACT. Distinct trajectories distinguish antigen-specific T cells in peanut-allergic individuals undergoing oral immunotherapy. J Allergy Clin Immunol. 2023 Jul;152(1):155-166.e9. doi: 10.1016/j.jaci.2023.03.020. Epub 2023 Mar 30. PMID 37003475
- [Background] Zhou X, Yu W, Lyu SC, Macaubas C, Bunning B, He Z, Mellins ED, Nadeau KC. A positive feedback loop reinforces the allergic immune response in human peanut allergy. J Exp Med. 2021 Jul 5;218(7):e20201793. doi: 10.1084/jem.20201793. Epub 2021 May 4. PMID 33944900
- [Background] Wanniang N, Boehm TM, Codreanu-Morel F, Divaret-Chauveau A, Assugeni I, Hilger C, Kuehn A. Immune signatures predicting the clinical outcome of peanut oral immunotherapy: where we stand. Front Allergy. 2023 Oct 2;4:1270344. doi: 10.3389/falgy.2023.1270344. eCollection 2023. PMID 37849958
- [Background] Neeland MR, Andorf S, Manohar M, Dunham D, Lyu SC, Dang TD, Peters RL, Perrett KP, Tang MLK, Saffery R, Koplin JJ, Nadeau KC. Mass cytometry reveals cellular fingerprint associated with IgE+ peanut tolerance and allergy in early life. Nat Commun. 2020 Feb 27;11(1):1091. doi: 10.1038/s41467-020-14919-4. PMID 32107388
- [Background] Sampson HA, Gerth van Wijk R, Bindslev-Jensen C, Sicherer S, Teuber SS, Burks AW, Dubois AE, Beyer K, Eigenmann PA, Spergel JM, Werfel T, Chinchilli VM. Standardizing double-blind, placebo-controlled oral food challenges: American Academy of Allergy, Asthma & Immunology-European Academy of Allergy and Clinical Immunology PRACTALL consensus report. J Allergy Clin Immunol. 2012 Dec;130(6):1260-74. doi: 10.1016/j.jaci.2012.10.017. No abstract available. PMID 23195525
- [Background] Pajno GB, Fernandez-Rivas M, Arasi S, Roberts G, Akdis CA, Alvaro-Lozano M, Beyer K, Bindslev-Jensen C, Burks W, Ebisawa M, Eigenmann P, Knol E, Nadeau KC, Poulsen LK, van Ree R, Santos AF, du Toit G, Dhami S, Nurmatov U, Boloh Y, Makela M, O'Mahony L, Papadopoulos N, Sackesen C, Agache I, Angier E, Halken S, Jutel M, Lau S, Pfaar O, Ryan D, Sturm G, Varga EM, van Wijk RG, Sheikh A, Muraro A; EAACI Allergen Immunotherapy Guidelines Group. EAACI Guidelines on allergen immunotherapy: IgE-mediated food allergy. Allergy. 2018 Apr;73(4):799-815. doi: 10.1111/all.13319. Epub 2017 Dec 5. PMID 29205393
- [Background] Schoos AM, Bullens D, Chawes BL, Costa J, De Vlieger L, DunnGalvin A, Epstein MM, Garssen J, Hilger C, Knipping K, Kuehn A, Mijakoski D, Munblit D, Nekliudov NA, Ozdemir C, Patient K, Peroni D, Stoleski S, Stylianou E, Tukalj M, Verhoeckx K, Zidarn M, van de Veen W. Immunological Outcomes of Allergen-Specific Immunotherapy in Food Allergy. Front Immunol. 2020 Nov 3;11:568598. doi: 10.3389/fimmu.2020.568598. eCollection 2020. PMID 33224138
- [Background] Zhang L, Chun Y, Arditi Z, Grishina G, Lo T, Wisotzkey K, Agashe C, Grishin A, Wang J, Sampson HA, Sicherer S, Berin MC, Bunyavanich S. Joint transcriptomic and cytometric study of children with peanut allergy reveals molecular and cellular cross talk in reaction thresholds. J Allergy Clin Immunol. 2024 Jun;153(6):1721-1728. doi: 10.1016/j.jaci.2023.12.028. Epub 2024 Jan 23. PMID 38272374
- [Background] Klueber J, Czolk R, Codreanu-Morel F, Montamat G, Revets D, Konstantinou M, Cosma A, Hunewald O, Skov PS, Ammerlaan W, Hilger C, Bindslev-Jensen C, Ollert M, Kuehn A. High-dimensional immune profiles correlate with phenotypes of peanut allergy during food-allergic reactions. Allergy. 2023 Apr;78(4):1020-1035. doi: 10.1111/all.15408. Epub 2022 Jun 24. PMID 35700055